CLINICAL TRIAL: NCT06069934
Title: Expanded Access Protocol (EAP) for Pridopidine in People With Amyotrophic Lateral Sclerosis (PL101-ALS501)
Brief Title: A Second Intermediate-Size Expanded Access Protocol (EAP) for Pridopidine in People With Amyotrophic Lateral Sclerosis (Pridopidine EAP 2)
Status: No longer available | Type: Expanded Access
Sponsor: Prilenia (Industry)
Collaborators: Massachusetts General Hospital (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: PL101-ALS501
Record Dates: First submitted 2023-09-27; First posted 2023-10-06 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Pridopidine; Lou Gehrig's disease; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Dementia; Dyskinesias; Movement Disorders; Heredodegenerative Disorders, Nervous System; Neurodegenerative Diseases; Cognition Disorders; Neurocognitive Disorders; Mental Disorders
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Dementia; Dyskinesias; Movement Disorders; Heredodegenerative Disorders, Nervous System; Neurodegenerative Diseases; Cognition Disorders; Neurocognitive Disorders; Mental Disorders | interventions — pridopidine

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Pridopidine — Pridopidine 45 mg hard gelatin capsules once daily p.o. (or via feeding tube)

SUMMARY:
Protocol PL101-ALS501: This EAP will provide access to pridopidine for up to 200 patients with ALS who are ineligible for clinical trials.

DETAILED DESCRIPTION:
ALS: Pridopidine will be given at a dose of 45 mg twice daily p.o. (or via feeding tube) over a 2-week up-titration period; followed by pridopidine 45 mg twice daily p.o. (or via feeding tube) for the remainder of the treatment period (through Week 104).

Each patient will be followed for 2 years with regularly scheduled visits. The screening and baseline visits will be performed in person; subsequent visits may occur in person or remotely. Recommended in-person visits will occur at Weeks 12, 52, 78, and end of treatment (Week 104 or early termination). If the patient is unable to complete the visits in person, these visits may also be completed remotely.

ELIGIBILITY:
Inclusion Criteria Amyotrophic Lateral Sclerosis (ALS):

* Sporadic or familial ALS.
* Patient does not qualify for clinical trials of pridopidine or as per site investigator's opinion, and is not medically or geographically suitable for other clinical trials.
* Capable of providing informed consent and complying with study procedures, in the site investigator's opinion.
* Patient has established care with a physician at a specialized ALS center involved in the study and will maintain this clinical care throughout the duration of the EAP.
* Pridopidine naive patients must have a life expectancy of at least 6 months in the site investigator's opinion.

Exclusion Criteria ALS:

* Confirmed prolonged Fridericia-corrected QT (QTcF) interval (>450 ms for men; >470 ms for women).
* Clinically significant heart disease, clinically significant history of arrhythmia, symptomatic or uncontrolled atrial fibrillation despite treatment, asymptomatic sustained ventricular tachycardia, or left bundle branch block.
* Known history of long QT syndrome or a first degree relative with long QT syndrome.
* Use of prohibited medications within the 4 weeks prior to baseline.
* Use of Nuedexta (>20 mg dextromethorphan and >10 mg quinidine twice daily); citalopram >20 mg/day; escitalopram >10 mg/day.
* Known allergy to pridopidine or any of the exipients (silicified microcrystalline cellulose, magnesium stearate).
* History of any clinically significant or unstable medical condition or laboratory abnormality that, based on site investigator's judgment, may interfere with assessment of the study objectives.
* Female who is pregnant or nursing or who plans to get pregnant during the course of the EAP.
* Female of child-bearing potential or male unwilling or unable to use accepted methods of birth control.
* Use of investigational treatments for ALS (as part of participation in a clinical trial or another EAP) within 5 half-lives (if known) or 30 days (whichever is longer) prior to screening (other than pridopidine).
* Patient receives or has received any gene or cell-based therapy.
* Active cancer or history of cancer, except for basal cell carcinoma or successfully treated squamous cell carcinoma of the skin, cervical carcinoma in situ, prostatic carcinoma in situ, or other malignancies curatively treated and with no evidence of disease recurrence for at least 3 years.
* Patients who chose to take experimental medications and/or supplements, and for whom this is the only reason they are not eligible for trials.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (32):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California, San Diego Health, La Jolla, California
  - UC Irvine, Orange, California
  - California Pacific Medical Center - Forbes Norris MDA/ALS Research Center, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - Nova Southeastern University, Fort Lauderdale, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Hospital Medical Center, Burlington, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Essentia Health, Duluth, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate, Syracuse, New York
  - Duke University, Durham, North Carolina
  - OhioHealth, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Lewis Katz School of Medicine at Temple University, Philadelphia, Pennsylvania
  - Texas Neurology, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- CHALS-CCT Program, UPR-MSC, San Juan, Puerto Rico